CLINICAL TRIAL: NCT02846467
Title: Comparison of Understanding of Informed Consent Between Portable Video Media Versus Written Consent at Urological Surgeries.
Brief Title: Information Improvement for Surgical Patients Through Portable Video Media
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Puerto Real (Other)
Collaborators: University of Cadiz (Other)
Responsible Party: Principal Investigator, Sebastian Armijos, PhD Urologist, Hospital Universitario Puerto Real
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HospitalUPR
Record Dates: First submitted 2016-07-22; First posted 2016-07-27 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Prostatic Hyperplasia; Bladder Cancer
Keywords: Informed consent; Patient Education; Mobile applications
MeSH Terms: conditions — Prostatic Hyperplasia; Urinary Bladder Neoplasms | interventions — Amyloid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Portable video media (Experimental): Patients who receive informed consent trough portable video media around 10 minutes
  Interventions: Other: Informed consent trough a portable video media
- Traditional IC (Active Comparator): Patients who receive traditional IC (written consent) during 10 to 15 minutes
  Interventions: Other: Written informed consent

INTERVENTIONS:
Other: Informed consent trough a portable video media — Information provided to patients using the mobile application (iURO app)
  Other Names: iURO Application (App)
  Arms: Portable video media
Other: Written informed consent — Information provided to patient trough the traditional informed consent (written IC) for transurethral resection of bladder or prostate.
  Other Names: Traditional informed consent; Standard verbal communication
  Arms: Traditional IC

SUMMARY:
The aim of this study is to evaluate the comprehension of the Informed consent with the Standard Verbal Communication (SVC) versus Portable Video Media (PVM).

DETAILED DESCRIPTION:
The informed consent (IC) is a fully ethical and legal consolidated requirement. IC is the voluntary authorization by a patient for surgical treatment (MeSH). The IC has to include: 1. What is and for what is it, 2. How is it made, 3. What effect will produce, 4. which patients will benefit, 5. Alternatives, 6. Risks and special situations.

The standard IC is based in written and verbal information, but the information provided is insufficient, leading to misunderstanding and even litigation.

Technology plays an important role in the improvement of IC: the portable video media, tablet, with the application (app) iURO assists the procedure through videos and illustrations.

To evaluate and measure the comprehension of the information that patients received, we elaborated and validated a "Questionnaire to evaluate the comprehension of IC" (the process was mounted as "Questionnaire for urology IC validation" in the poster session at the 17th International European Association of Urology Nurses (EAUN) Meeting, Munich-Germany).

The patients undergoing to bladder or prostate transurethral resection were selected. Afterwards they were randomized previous the interview, into two groups: patients informed by PVM with the app iUro (experimental group) versus patients with an SVC (control group). The questionnaire was used to compare the comprehension of the surgery immediately and 15 days after the surgery. The items regarding questionnaire were: information, utility of the intervention, side effects, complications, comorbidity, usefulness of information, anxiety and risks.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are going to receive transurethral resection of bladder or prostate
* Patients, women and men, older than 18 years without any mental disability

Exclusion Criteria:

* Patients who refuse to participate in the study
* Patients who have inability to communicate in spanish.
* Several visual problems that limit the ability to read written material

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2013-12; Primary Completion 2015-10 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Comprehension of informed consent | Prior to surgery

SECONDARY OUTCOMES:
Comprehension of informed consent | 15 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Armijos Leon, Urologist, Principal Investigator — Hospital Universitario Puerto Real; Federico Rodriguez Rubio, Urologist, Study Director — Univesity of Cadiz; Jorge Rioja Zuazu, Urologist, Study Chair — Universidad de Zaragoza
Locations (1):
- Urology Department of the University Hospital of Puerto Real, Puerto Real, Cadiz, Spain

IPD SHARING:
Plan to Share IPD: Yes
The database with the demographic and results of the participant is going to be available during the next six months. The information will be send with an email request.

REFERENCES:
- See also: Abstract entitled: "MHealth (Mobile Health):The use of portable video media versus standard verbal communication in the informed consent", presented at 5th Meeting of Uro-Technology (ESUT) held in Athens, Greece — https://twitter.com/Uroweb/status/752027133837471744/photo/1